CLINICAL TRIAL: NCT03140462
Title: The Influence of ABCB1、CYP3A4、CYP3A5、POR Genetic Polymorphism of Donor on Tacrolimus Blood Concentration in Liver Transplant Patients
Brief Title: Influence of Genetic Polymorphism of Donor on Tacrolimus Concentration in Liver Transplant
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201612023RIND
Record Dates: First submitted 2017-04-24; First posted 2017-05-04 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2020-12

CONDITIONS: Liver Transplantation
Keywords: Tacrolimus; Pharmacokinetics; Genetic polymorphisms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood , paraffin-embedded liver biopsy, or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- liver transplant patients and donors: To study clinical and genetic factors on tacrolimus dose normalized trough concentration.

SUMMARY:
To study the influence of donor's ABCB1、CYP3A4、CYP3A5、POR genetic polymorphism on tacrolimus blood concentration in liver transplant recipients.

DETAILED DESCRIPTION:
This study will start with a retrospective data analysis. The investigators will use the electronic databases of National Taiwan University Hospital to identify patients who underwent liver transplantation, received tacrolimus and were still followed up at the outpatient clinic. Inclusion and exclusion criteria will be applied to screen appropriate participants, and find their donors. And analyze the effect of genetic polymorphism (ABCB1、CYP3A4、CYP3A5、POR) of donors, including other factors of recipients, on the dose normalized trough concentration of tacrolimus.

ELIGIBILITY:
Inclusion Criteria:donors' recipients

* Living liver transplant during 20070101 ~ 20151231 and only received liver transplantation
* Lab data at least 8 months,
* Receiving tacrolimus as immunosuppressive drugs
* Transplantation at 20 ~ 65 years old

Exclusion Criteria: donors' recipients

* Retransplantation or multi-organ transplantation
* Non-Asian
* Positive for human immunodeficiency virus.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplant patients' donors
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-05-21 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Dose normalized trough concentration of tacrolimus in liver transplant patients within the first 6 months post-transplantation | Within the first 6 months post-transplantation
  Analyse the effect of the donor's genetic polymorphism to dose normalized trough concentration of tacrolimus in liver transplant patients. Trough level of tacrolimus was adjusted by liver recipient's body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Rey-Heng Hu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No